CLINICAL TRIAL: NCT06756451
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of RJK-RT2831 Injection in Patients With Hematologic Malignancies.
Brief Title: This Study is a FIH Study Which is Required to Understand the PK Characteristics, MTD, RP2D and Safety Profile.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing RegeneCore Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJK-RT2831-101
Record Dates: First submitted 2024-11-27; First posted 2025-01-03 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Malignancies
Keywords: RT-RT2831; Malignancies
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RJK-RT2831 (Experimental)
  Interventions: Drug: RJK-RT2831 dose-escalation phase Ia; Drug: RJK-RT2831 Dose Expansion Phase Ib

INTERVENTIONS:
Drug: RJK-RT2831 dose-escalation phase Ia — there are seven doses(1mg-160mg) in this part. The subjects will receive RJK-RT2831 injection twice a week by intravenous push or intravenous infusion for 4 weeks until the end of one dosing cycle (28 days). After one dosing cycle, if the subject tolerates, the subject will continue to receive treatment until the researcher believes that the subject no longer benefits, or the subject has disease progression, unacceptable toxicity, withdraws informed consent, dies, is lost to follow-up, or starts new anti-tumor treatment (whichever occurs first).
Drug: RJK-RT2831 Dose Expansion Phase Ib — there are four doses in this part. The subjects will be randomized in a 1:1 ratio to receive one dose level of RJK-RT2831 intravenous infusion twice a week for 4 weeks until the end of one dosing cycle (28 days).After one dosing cycle, if the subject tolerates, the subject will continue to receive treatment until the researcher believes that the subject no longer benefits, or the subject has disease progression, unacceptable toxicity, withdraws informed consent, dies, is lost to follow-up, or starts new anti-tumor treatment (whichever occurs first).

SUMMARY:
This study is a first-in-human (FIH) study which is required to understand the safety, tolerability, pharmacokinetics and preliminary efficacy of RJK-RT2831 injection in patients with hematologic malignancies

DETAILED DESCRIPTION:
This is the first-in-human, Phase 1, open-label, multicenter, dose-escalation and dose expansion phase study to investigate the safety, Tolerability, pharmacokinetics and preliminary efficacy of RJK-RT2831 injection in patients with hematologic malignancies. About 70 subjects with malignant blood tumors will be recruited. The specific tumor type will be determined based on the results of the Phase Ia trial and may be expanded to other malignant blood tumor types.The primary goal of the study is to assess the safety, tolerability, maximum tolerated dose (MTD),determine the recommended doses for expansion (RDEs) and recommended phase 2 dose (RP2D) in patients with hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* 1. A male or female aged ≥ 18 and <75 years old.
* 2. The following three points are evaluated by the investigator and are deemed suitable to participate in the study: a) The subject fully understands the requirements of this study and voluntarily signs a written informed consent form; b) Be able to comply with the medication requirements of this study as well as all study related procedures and assessments; c) Not deemed as potentially unreliable and/or uncooperative.
* 3. An ECOG physical status score is ≤ 2 and an expected survival is ≥ 3 months.
* 4. Relapsed or refractory acute myeloid leukemia (AML) that meets the following criteria will be included in Phase Ⅰa : Patients diagnosed with AML according to the 5th edition of the World Health Organization (WHO) Classification of Haematolymphoid Tumours: -Myeloid and Histiocytic/Dendritic Neoplasms (Khoury et al., 2022), including any subtype except for acute promyelocytic leukemia (APL). These patients must have received at least one previous treatment and have failed to current standard treatments that provide clinical benefit.

Note: The following diagnostic criteria must be met for relapsed/refractory AML: (1) Relapsed AML: Leukemia cells reappear in the peripheral blood or bone marrow blast cells exceed 5% after complete remission (CR) (excluding reasons such as bone marrow regeneration post-consolidation chemotherapy) or there is extramedullary infiltration by leukemia cells. (2) Refractory AML: Initial cases that are unresponsive after two cycles of standard regimen treatment; recurrence within 12 months after CR and consolidation therapy; recurrence beyond 12 months with ineffectiveness of conventional chemotherapy; those who have relapsed twice or more; or persistent extramedullary leukemia.;

-5. Phase Ib tentatively includes patients with hematologic malignancies that meet the following criteria: relapsed or refractory AML subjects who have received at least one previous treatment and have failed to current standard treatments that provide clinical benefit, and MDS subjects who are diagnosed according to the 5th edition of the WHO Classification of Haematolymphoid Tumours-Myeloid and Histiocytic/Dendritic Neoplasms (Khoury et al., 2022) and are classified as high-risk or very-high-risk according to the Revised International Prognostic Scoring System (IPSS-R) (Greenberg et al., 2012). The specific tumor type will be determined based on the results of the Phase Ia trial and may be extended to other hematologic malignancies.

Note: Subjects with myelodysplastic syndromes with excess blasts (MDS-EBs) type 1 (MDS-EB1) or type 2 (MDS-EB2) may be considered for inclusion. The EB type has a higher risk of transformation to AML than other subtypes and may have greater clinical benefits.

* 6. The test of CD33 and/or CD123 for Phase Ia and Ib subjects in this study will be required to be positive, and patients with any level of CD33 and/or CD123 positivity were allowed to be included. Note: The positivity and expression levels of CD33 and CD123 were determined by each site.
* 7. Consent to bone marrow biopsy and aspiration, and consent to implantation of medical devices such as peripherally inserted central catheter (PICC), or venous access port, or central venous catheter (CVC) (if applicable) for long-term intravenous drug administration.
* 8. Patients have recovered from toxicity of prior first-line therapy, i.e., Grade 1 toxicity according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) V5.0, with the exception of toxicities such as alopecia, fatigue, and other toxicities deemed by the investigator to be of no safety risk to the patient, as well as hematological toxicities related to the tumor.
* 9. Substantial normal function of major organs with screening laboratory tests meeting the following criteria:

  1. Bone marrow function: white blood cell count ≤ 30×10^9/L;
  2. Liver function: TBIL ≤ 1.5×ULN, TBIL ≤ 3×ULN if Gilbert's syndrome; ALT and AST ≤ 3 ×ULN;
  3. Renal function: creatinine clearance rate (CCr) > 50 mL/min calculated according to the Cockcroft-Gault method
  4. Coagulation function: activated partial thromboplastin time (APTT) and prothrombin time (PT) ≤ 1.5×ULN.
* 10. The serum pregnancy test for female patients of childbearing potential should be negative during the screening period. Male and female patients of childbearing potential must agree to use effective methods of contraception from signing an informed consent form during the screening period, throughout the study and for 3 months after the last dose of the RJK-RT2831, including but not limited to: abstinence, vasectomy in males, female sterilization surgery, effective intrauterine contraceptive devices or condoms, and effective contraceptive medications.. Note: Women of non-childbearing potential include permanent infertility (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) and postmenopausal women.

Exclusion Criteria:

* 1. APL is suspected or confirmed based on morphology, immunophenotyping, molecular testing, or chromosomal karyotyping, or other hematological tumors, such as myeloid sarcoma, mixed phenotype acute leukemia, accelerated phase and blast phase of chronic myeloid leukemia, etc.;
* 2. Has received any anticancer therapy or investigational drug within the following specified time period prior to the first dose of RJK-RT2831:

  1. Received cytotoxic chemotherapy (except hydroxyurea use for subjects with leukocytosis >10,000 cells/mm3 or rapid disease progression), radiotherapy (except local palliative radiotherapy), immunotherapy, targeted therapy and other anti-tumor treatments within 14 days;
  2. Received adoptive cell therapy, such as autologous or donor natural killer cell or T lymphocyte infusions (e.g., chimeric antigen receptor-T cells), unless > 60 days prior to the first dose of study treatment and treatment-related toxicities have resolved to at least Grade 1;
  3. Received any investigational drug (for any indication) within 5 half-lives of the drug or 14 days, whichever is longer;
  4. Received an autologous haematopoietic stem cell transplant within 12 weeks.
* 3. Subjects with cardiovascular disease, including but not limited to:

  1. Resting state, mean QTcF > 480 ms in men/women derived from 12-lead electrocardiogram (ECG) (repeated 3 times); Note: QTcF = QTcB ×RR^0.17, QTcB is the corrected QT interval obtained using the Bazetts correction formula;
  2. Echocardiogram or multigated acquisition (MUGA) scan showing a left ventricular ejection fraction of less than 50%;
  3. Symptomatic or treatment-requiring abnormalities in rhythm, conduction, and resting ECG morphology, such as arrhythmias, degree II or III atrioventricular block, congestive heart failure (New York Heart Association cardiac function class III or IV)
  4. New onset of angina pectoris and myocardial infarction within 6 months prior to initiation of study treatment;
  5. Various factors that may increase the risk of prolonged QTc, such as congenital long QT syndrome, having long QT syndrome in the immediate family history, and being on any medications known to prolong the QT interval.
  6. History of cerebral perfusion (e.g., carotid artery stenosis) or stroke or transient ischemic attack within 6 months prior to screening.
* 4. Subjects with an evidence of infectious disease, including:

  1. Hepatitis B surface antigen (HBs Ag) positive, and hepatitis B virus deoxyribonucleic acid (HBV DNA) copy number greater than the normal upper limit;
  2. Hepatitis C virus antibody (HCV Ab) positive and hepatitis C virus ribonucleic acid (HCV RNA) levels greater than the normal upper limit;
  3. infected with human immunodeficiency virus (HIV);
  4. Treponema pallidum (Tp) antibody positive;
  5. Known active tuberculosis.
* 5. Subjects with leukemic extramedullary infiltration.
* 6. Subjects with long-term steroid therapy, except for the following: 10 mg of prednisone daily (or equivalent) or lower dose steroids for the control of nausea, vomiting, seasonal allergies, or for the prevention of adrenocortical insufficiency. Subjects who require > 10 mg of prednisone for a long time (e.g., more than 2 months) need to be excluded.Note: Topical steroids or inhaled steroids are permitted.
* 7. Subjects with autoimmune hemocytopenia that the investigator assessed as requiring active intervention, e.g. autoimmune haemolytic anaemia, idiopathic thrombocytopenic purpura.
* 8. Subjects who have undergone major surgical procedures (craniotomy, thoracotomy, laparotomy, vascular intervention, other as defined by the investigator) or have unhealed wounds, ulcers or fractures within 4 weeks prior to the first dose of RJK-RT2831. Note: For palliative care purposes, local surgical treatment of isolated lesions is acceptable.
* 9. Subjects with uncontrolled co-morbidities such as:

  1. Severe infection, including but not limited to hospitalization due to infection, bacteremia, or severe pneumonia complications, occurs within 4 weeks prior to initiation of study treatment; or patients who have received therapeutic oral or intravenous antibiotics within two weeks prior to starting study treatment, except who have received prophylactic antibiotics (e.g., for the prevention of urinary tract infection or chronic obstructive pulmonary disease). If it is not an active infection and the infection is controllable, the subjects can be enrolled;
  2. Other malignancies (other than non-melanoma basal cell carcinoma or squamous cell carcinoma of the skin, breast/cervical carcinoma in situ, superficial bladder carcinoma that have received radical treatment and no evidence of disease recurrence) within 5 years prior to initiation of RJK-RT2831 treatment or concurrently;
  3. Subjects with current cancerous meningitis, spinal cord compression, etc.;
  4. A history of poorly controlled hypertension (abnormal blood pressure measured 3 times to take the mean, systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg);
  5. Other acute or chronic illnesses or abnormal laboratory test values that may result in an increase in the risk associated with study participation or investigational drug administration, or interfere with the interpretation of study results;
* 10. Subjects who are expected to receive other anti-tumor therapy during the study (palliative radiotherapy is allowed).
* 11. Subjects with prior therapy using gemtuzumab ozogamicin or other CD33-targeting agents, or who have experience with CD33-targeting compounds in the clinical trial phase.
* 12.Subjects with prior therapy using tagraxofusp or other CD123-targeting agents, or who have experience with CD123-targeting compounds in the clinical trial phase.
* 13.Subjects who are allergic to prescription components of the RJK-RT2831 formulation (histidine, histidine hydrochloride, sucrose, Poloxam 188).
* 14.Subjects who are pregnant or lactating women.
* 15.Subjects who have received other investigational drugs within 2 cycles prior to medication, or are concurrently participating in another interventional clinical study (unless they are participating in an observational study or are in the follow-up phase of an interventional study).
* 16.Subjects with a previous history of receiving allogeneic organ transplantation and allogeneic haematopoietic stem cell transplantation.
* 17. In the opinion of the investigator, the subject has other factors that may affect the results of the study and interfere with his/her participation throughout the study, including previous or existing medical conditions, laboratory abnormalities, and the subject's unwillingness to comply with the processes, restrictions, and requirements of the study.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2028-04-08 (Estimated); Study Completion 2028-07-14 (Estimated)

PRIMARY OUTCOMES:
phase Ia and phase Ib: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | The summary of all AEs was dominated by adverse events that occurred during treatment, including any AE that occurred from the first administration of the study drug until 28 ± 7 days after the last administration.
  All AEs (except for CRS and TLS) will be graded according to NCI CTCAE V5.0, a common standard term for AE.
  CRS and TLS will be graded according to ASCTC Consensus (2019) and Cairo-Bishop grading system (Howard revised) respectively.
phase Ia: Maximum Tolerated Dose (MTD) | From the first administration of the study drug until 28 days after the first dose
  To assess the safety, tolerability, and maximum tolerated dose (MTD) of RJK-RT2831 in patients with hematologic malignancies.
phase Ia: Recommended Doses for Expansion (RDEs) | From the first administration of the study drug until 28 ±7 days after the last administration and prior to the initiation of a new anti-tumor therapy
  To determine the recommended doses for expansion (RDEs) in patients with hematologic malignancies.
phase Ib: Recommended Phase II Dose (RP2D) | From the first administration of the study drug until 28 ±7 days after the last administration and prior to the initiation of a new anti-tumor therapy
  To determine the recommended Phase II dose (RP2D) in patients with hematologic malignancies.

SECONDARY OUTCOMES:
Cmax | The first 6 cycles (28 days/cycle)
  Pharmacokinetic (PK) analysis of RT2831
Tmax | The first 6 cycles (28 days/cycle)
  PK analysis of RT2831
Area under the concentration-time curve (AUC) | The first 6 cycles (28 days/cycle)
  PK analysis of RT2831
Total Clearance (CL) | The first 6 cycles (28 days/cycle)
  PK analysis of RT2831
Volume of distribution (Vd) | The first 6 cycles (28 days/cycle)
  PK analysis of RT2831
Half-life (t1/2) | The first 6 cycles (28 days/cycle)
  PK analysis of RT2831
Clearance (CL) | The first 6 cycles (28 days/cycle)
  PK analysis of RT2831
volume of distribution (Vd） | The first 6 cycles (28 days/cycle)
  PK analysis of RT2831
elimination rate constant (Kel) | The first 6 cycles (28 days/cycle)
  PK analysis of RT2831
average concentration (Cave) | The first 6 cycles (28 days/cycle)
  PK analysis of RT2831
Anti-Drug Antibodies (ADA) | On the first day of each cycle until the last cycle administrated (28 days/cycle)
  Monitor the production of anti-drug antibodies (ADA) during the dose escalation and dose expansion phases.
overall remission rate (ORR) | On the first day of each cycle until the end of treatment (+ 3 days) and before starting new anti-tumor therapy (28 days/cycle)
  Includes: complete remission (CR), complete remission with incomplete blood count recovery (CRi), partial remission (PR)
duration of remission (DOR) | Throughout the study (from the first administration of the study drug until 28 ± 7 days after the last dose and before starting new anti-tumor therapy)
  DOR is calculated from date of initial documentation of a response (complete response (CR) and complete remission with incomplete blood count recovery (CRi) or partial response (PR) to the date of first documented evidence of relapse, defined in disease-specific response criteria, or death, whichever occurs first.
event-free survival (EFS) | Throughout the study (until 28 ± 7 days after the last dose and before starting new anti-tumor therapy)
  time from the date of first study treatment administration to the date of treatment failure, hematologic relapse from CR/CRi/PR or death from any cause
overall survival (OS) | Throughout the study (every 3 months ±7 days after discontinuation to assess survival status until subject death or study termination)
  time from the date of first study treatment administration to the date of death

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - The First Affiliated Hospital of USTC, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Tangshan Central Hospital, Tangshan, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No